CLINICAL TRIAL: NCT07378579
Title: A Phase 1, Partially Blinded, Randomized, Crossover Study to Evaluate the Pharmacokinetics and QT/QTc Interval of ESK-001 Compared to Placebo and Moxifloxacin in Healthy Subjects
Brief Title: An Investigational Study to Evaluate the Cardiac Safety Assessment (TQTc Study) of ESK-001
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alumis Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: ESK-001-019
Record Dates: First submitted 2025-12-10; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: All subjects will be randomized to 1 of 4 treatment sequences; each subject will receive all 4 treatments. Treatments 1 through 3 will be blinded; Treatment 4 will be given open label. The central ECG laboratory will be blinded to treatment assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Treatment 1: (Therapeutic dose) (Experimental): 1 oral dose of ESK-001
  Interventions: Drug: ESK-001
- Treatment 2: (Supratherapeutic dose) (Experimental): 1 oral dose of ESK-001
  Interventions: Drug: ESK-001
- Treatment 3: ESK-001-matched placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Treatment 4: (positive control) (Active Comparator): Moxifloxacin 400 mg tablet
  Interventions: Drug: Moxifloxacin (400 mg)

INTERVENTIONS:
Drug: ESK-001 — Single oral dose of ESK-001 in participants
  Arms: Treatment 1: (Therapeutic dose); Treatment 2: (Supratherapeutic dose)
Drug: Moxifloxacin (400 mg) — positive control
  Arms: Treatment 4: (positive control)
Drug: Placebo — ESK-001-matched placebo
  Arms: Treatment 3: ESK-001-matched placebo

SUMMARY:
This a phase 1, partially blinded, randomized, crossover study to determine the pharmacokinetics (PK) and QT/QTc interval of study drug (ESK-001) in healthy volunteer participants,

DETAILED DESCRIPTION:
This clinical trial information was submitted voluntarily under the applicable law and, therefore, certain submission deadlines may not apply. (That is, clinical trial information for this applicable clinical trial was submitted under section 402(j)(4) (A) of the Public Health Service Act and 42 CFR 11.60 and is not subject to the deadlines established by sections 402(j)(2) and (3) of the Public Health Service Act or 42 CFR 11.24 and 11.44.)

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects aged between 18 and 55 years, inclusive. Body mass index between ≥18.0 and ≤32.0 kg/m2, inclusive, and a minimum body weight of 45 kg.
* Able to comprehend and willing to sign an ICF and to abide by the study restrictions.
* In good health, determined by no clinically significant findings from medical history, 12-lead ECG, vital signs measurements, and clinical laboratory evaluations, and from the physical examination at screening or check-in, as assessed by the investigator (or designee).
* Serum sodium, potassium, calcium, and magnesium levels are within the normal range at screening and check-in-

Exclusion Criteria:

* Positive hepatitis panel and/or positive human immunodeficiency virus test, hepatitis B surface antigen, or hepatitis C antibodies.
* Alanine aminotransferase or aspartate aminotransferase >1.5 times the upper limit of normal, at screening or check-in.
* History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, as determined by the investigator (or designee).
* Surgery within the past three months prior to the first study drug administration determined by the principal investigator to be clinically relevant.
* History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs (uncomplicated appendectomy and hernia repair are allowed).
* History of Gilbert's syndrome or cholecystectomy surgery.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2024-06-21 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline in placebo-adjusted QTcF (∆∆QTcF) | 24 hours

SECONDARY OUTCOMES:
Change from baseline in ECG parameter ΔHR | 24 hours
Change from baseline in ECG parameter Δ PR interval | 24 hours
Change from baseline in ECG parameter ΔQRS duration | 24 hours
Change from baseline in ECG parameter ΔQTc interval | 24 hours
Incidence of nonserious adverse events (AE), serious adverse events (SAE), and AE leading to discontinuation | Up to 22 Days
Number of clinically significant changes in clinical laboratory values, vital signs, ECGs, and physical examinations | Up to 22 Days
Composite of pharmacokinetic (PK) parameter Vz/F for ESK-001 and metabolites | 24 hours
Composite of pharmacokinetic (PK) parameter Cmax for ESK-001 and metabolites | 24 hours
Composite of pharmacokinetic (PK) parameter tmax for ESK-001 and metabolites | 24 hours
Composite of pharmacokinetic (PK) parameter CL/F for ESK-001 and metabolites | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Jorn Drappa, MD, Ph.D., Study Director — Alumis Inc
Locations (1):
- Fortrea CRU, Daytona Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided
The Sponsor Alumis Inc. is a clinical-stage pharmaceutical company that has not yet adopted an Individual Participant Data (IPD) sharing plan.